CLINICAL TRIAL: NCT03125200
Title: A Phase 1, Open-Label, Dose-Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Antitumor Activity of ADCT-502 in Patients With Advanced Solid Tumors With HER2 Expression
Brief Title: Study of ADCT-502 in Patients With Advanced Solid Tumors Withhuman Epidermal Growth Factor Receptor-2 (HER2) Expression
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Safety
Sponsor: ADC Therapeutics S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADCT-502-101
Record Dates: First submitted 2017-04-10; First posted 2017-04-24 (Actual); Results first posted 2019-08-28 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Breast Cancer; Non Small Cell Lung Cancer; GastroEsophageal Cancer; Bladder Cancer
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ADCT-502 (Experimental): Part 1 (dose escalation): Participants received an infusion of ADCT-502, at escalating doses. Part 1 continued until the maximum tolerated dose or the recommended dose(s) and schedule(s) for expansion were determined.
  Part 2 (expansion): Participants were due to be assigned to the recommended dose level of ADCT-502 as identified in Part 1 by the Dose Escalation Steering Committee.
  Interventions: Drug: ADCT-502

INTERVENTIONS:
Drug: ADCT-502 — Intravenous Infusion

SUMMARY:
This study evaluated ADCT-502 in participants with Advanced Solid Tumors with HER2 Expression. Participants participated in a dose-escalation phase (Part 1) and were due to participate in the dose expansion phase (Part 2). In Part 2, patients were due to receive the dose level identified in Part 1, but the study was terminated prior to the beginning of Part 2.

DETAILED DESCRIPTION:
Study ADCT-502-101 was the first clinical study with ADCT-502 in participants with Advanced Solid Tumors with HER2 Expression.

ADCT-502 is an antibody drug conjugate (ADC) composed of an engineered version of the humanized monoclonal antibody trastuzumab, directed against the human HER2 receptor, conjugated to a pyrrolobenzodiazepine (PBD) dimer cytotoxin. ADCT-502 specifically binds to HER2, and once internalized, releases the PBD dimer to allow cross-linking of DNA and eventually trigger cell death.

The study had 2 parts. In Part 1 (dose escalation) participants received an infusion of ADCT-502, at escalating doses. Part 1 continued until the maximum tolerated dose or the recommended dose(s) and schedule(s) for expansion were determined. In Part 2 (expansion), participants were due to be assigned to the recommended dose level of ADCT-502 identified in Part 1 by the Dose Escalation Steering Committee, but the study was terminated prior to the beginning of Part 2.

For each participant, the study included a screening period (up to 28 days), a treatment period, and a follow-up period to assess disease progression and survival for up to 12 weeks after the last dose of study drug. The total study duration was dependent on overall participant tolerability to the study drug and response to treatment as participants were able to continue treatment until disease progression or unacceptable toxicity.

ELIGIBILITY:
Main Inclusion Criteria:

* Male or female age 18 years or older
* Refractory to or intolerant of existing therapy(ies) known to provide clinical benefit for their condition.
* Eastern Cooperative Oncology Group (ECOG) performance status: Part 1: 0-2, Part 2: 0-1
* Availability of formalin-fixed paraffin-embedded (FFPE) tumor tissue block or unstained slides to demonstrate HER2 expression.
* Pathologic diagnosis of solid tumor malignancy that is locally advanced or metastatic at time of Screening with documented HER2 expression.
* Part 2/Dose Expansion Only: Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
* Absolute neutrophil count (ANC) ≥ 1500/mm3 (≥1.5× 109/L).
* Platelet count ≥100,000 //mm3 (≥100 × 109/L).
* Hemoglobin ≥ 9 g/L (≥5.6 mmol/L).
* Aspartate transaminase (AST) and alanine aminotransferase (ALT) ≤ 2.5 x upper limit of normal (ULN); or ≤ 5.0 × ULN if liver metastases are present.
* Total bilirubin ≤ 1.5× ULN (or ≤ 3× ULN, with direct bilirubin ≤1.5 × ULN, in participants with known Gilbert syndrome).
* Creatinine ≤ 1.5× ULN; or, if serum creatinine > 1.5 × ULN, a measured creatinine clearance must be >60mL/min/1.73m2 as calculated by the Cockcroft and Gault equation for participants to be eligible.
* Women of childbearing potential must agree to use a highly effective method of contraception from the time of giving informed consent until at least 16 weeks after the last dose of ADCT-502. Men with female partners who are of childbearing potential must agree that they or their partners will use a highly effective method of contraception from the time of giving informed consent until at least 16 weeks after the participant receives his last dose of ADCT-502.

Main Exclusion Criteria:

* Known history of ≥ Grade 3 hypersensitivity to a therapeutic antibody.
* Known history of positive serum human anti-drug antibody (ADA) to trastuzumab.
* Major surgical procedure or significant traumatic injury, radiotherapy, chemotherapy, targeted therapy, hormone therapy, or other anticancer therapy.
* Failure to recover to Grade 0 or Grade 1 from acute non-hematologic toxicity due to previous therapy, prior to screening (with the exception of alopecia).
* Central Nervous System (CNS) disease only.
* Symptomatic CNS metastases or evidence of leptomeningeal disease.
* Active cardiovascular disease or significant history thereof.
* Other active disease including but not limited to ulceration of the upper gastrointestinal tract, autoimmune disease, HIV infection, active Hepatitis B virus (HBV) and hepatitis C virus (HCV) infection.
* Breastfeeding or pregnant.
* Other concurrent severe and/or uncontrolled medical conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2018-04-05 (Actual); Study Completion 2018-04-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (4):
  - Stanford Cancer Center, Palo Alto, California
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering Memorial Hospital, New York, New York
  - South Texas Accelerated Research Therapeutics, LLC, San Antonio, Texas
- Medical Oncology Clinic - Institut Jules Bordet, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1: Dose 30μg/kg: Dose-escalation part of the study. Participants received ADCT-502 (30 μg/kg) via a 1-hour intravenous infusion once every 3 weeks.
- Part 1: Dose 60μg/kg: Dose-escalation part of the study. Participants received ADCT-502 (60 μg/kg) via a 1-hour intravenous infusion once every 3 weeks.
- Part 1: Dose 120μg/kg; Part 1: Dose 150μg/kg; Part 1: Dose 180μg/kg; Part 1: Dose 210μg/kg; Part 1: Dose 240μg/kg: Dose-escalation part of the study. Participants received ADCT-502 (120 μg/kg) via a 1-hour intravenous infusion once every 3 weeks.
Period: Overall Study
Arm/Group | Part 1: Dose 30μg/kg | Part 1: Dose 60μg/kg | Part 1: Dose 120μg/kg | Part 1: Dose 150μg/kg | Part 1: Dose 180μg/kg | Part 1: Dose 210μg/kg | Part 1: Dose 240μg/kg
Started | 2 | 2 | 2 | 5 | 4 | 3 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 2 | 2 | 5 | 4 | 3 | 3
Not completed — Study Termination | 0 | 0 | 0 | 1 | 1 | 2 | 1
Not completed — Clinical Progression | 0 | 0 | 0 | 1 | 0 | 1 | 0
Not completed — Progressive Disease | 2 | 1 | 2 | 1 | 2 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Toxicity | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Consent Withdrawn by Subject | 0 | 1 | 0 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Part 1: Dose 150μg/kg: Dose-escalation part of the study. Participants received ADCT-502 (150 μg/kg) via a 1-hour intravenous infusion once every 3 weeks.
- Part 1: Dose 180μg/kg: Dose-escalation part of the study. Participants received ADCT-502 (180 μg/kg) via a 1-hour intravenous infusion once every 3 weeks.
- Part 1: Dose 210μg/kg: Dose-escalation part of the study. Participants received ADCT-502 (210 μg/kg) via a 1-hour intravenous infusion once every 3 weeks.
- Part 1: Dose 240μg/kg: Dose-escalation part of the study. Participants received ADCT-502 (240 μg/kg) via a 1-hour intravenous infusion once every 3 weeks.
- Total: Total of all reporting groups
Arm/Group | Part 1: Dose 30μg/kg | Part 1: Dose 60μg/kg | Part 1: Dose 120μg/kg | Part 1: Dose 150μg/kg | Part 1: Dose 180μg/kg | Part 1: Dose 210μg/kg | Part 1: Dose 240μg/kg | Total
Number analyzed (Participants) | 2 | 2 | 2 | 5 | 4 | 3 | 3 | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 1 | 3 | 3 | 2 | 2 | 13
  >=65 years | 1 | 1 | 1 | 2 | 1 | 1 | 1 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 4 | 3 | 1 | 2 | 15
  Male | 1 | 0 | 0 | 1 | 1 | 2 | 1 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 1 | 2 | 2 | 5 | 4 | 3 | 3 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 2 | 1 | 2 | 3 | 4 | 3 | 2 | 17
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Belgium | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 3
  United States | 2 | 2 | 2 | 4 | 3 | 2 | 3 | 18
Height [Mean (Standard Deviation); unit: Centimetres] | 164.60 (7.920) | 161.00 (7.071) | 165.65 (1.909) | 161.02 (7.814) | 167.38 (9.571) | 169.33 (9.504) | 154.13 (11.055) | 163.21 (8.772)
Weight [Mean (Standard Deviation); unit: Kilograms] | 66.75 (6.576) | 76.85 (49.427) | 73.65 (21.850) | 61.70 (9.113) | 84.25 (22.422) | 67.93 (2.173) | 59.90 (10.300) | 69.69 (18.222)
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 24.61 (0.059) | 28.89 (16.514) | 26.94 (8.583) | 23.70 (2.218) | 30.33 (8.873) | 23.89 (3.330) | 25.13 (2.762) | 26.03 (6.241)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Dose-Limiting Toxicities
Time Frame: Day 1 to 3 Weeks (one cycle)
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Dose 30μg/kg | Part 1: Dose 60μg/kg | Part 1: Dose 120μg/kg | Part 1: Dose 150μg/kg | Part 1: Dose 180μg/kg | Part 1: Dose 210μg/kg | Part 1: Dose 240μg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 5 | 4 | 3 | 3
Participants | 0 | 0 | 0 | 0 | 1 | 0 | 1

2. Primary Outcome: Number of Participants Who Experienced a Dose-Limiting Toxicity With a CTCAE Grade of 3 or Above
Description: The Common Terminology Criteria For Adverse Events (CTCAE) Version 4 will be used.
Time Frame: Day 1 to 3 Weeks (one cycle)
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Dose 30μg/kg | Part 1: Dose 60μg/kg | Part 1: Dose 120μg/kg | Part 1: Dose 150μg/kg | Part 1: Dose 180μg/kg | Part 1: Dose 210μg/kg | Part 1: Dose 240μg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 5 | 4 | 3 | 3
Participants | 0 | 0 | 0 | 0 | 1 | 0 | 1

3. Primary Outcome: Number of Participants Who Experience At Least One Treatment Emergent Adverse Event (TEAE)
Description: An adverse event is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. A TEAE is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: Day 1 to end of trial, a maximum of 168 days (+ 30 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Dose 30μg/kg | Part 1: Dose 60μg/kg | Part 1: Dose 120μg/kg | Part 1: Dose 150μg/kg | Part 1: Dose 180μg/kg | Part 1: Dose 210μg/kg | Part 1: Dose 240μg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 5 | 4 | 3 | 3
Participants | 2 | 2 | 2 | 5 | 4 | 3 | 3

4. Primary Outcome: Number of Participants Who Experience At Least One Treatment Emergent Serious Adverse Event (SAE)
Time Frame: Day 1 to end of trial, a maximum of 168 days (+ 30 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Dose 30μg/kg | Part 1: Dose 60μg/kg | Part 1: Dose 120μg/kg | Part 1: Dose 150μg/kg | Part 1: Dose 180μg/kg | Part 1: Dose 210μg/kg | Part 1: Dose 240μg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 5 | 4 | 3 | 3
Participants | 0 | 1 | 0 | 2 | 1 | 2 | 1

5. Primary Outcome: Number of Participants With Clinically Significant Clinical Laboratory Tests
Description: Clinical significance was determined by the investigator.
Time Frame: Day 1 to end of trial, a maximum of 168 days (+ 30 days)
Population: This analysis was planned but data was not collected as the study was terminated due to safety reasons.
Arm/Group | Part 1: Dose 30μg/kg | Part 1: Dose 60μg/kg | Part 1: Dose 120μg/kg | Part 1: Dose 150μg/kg | Part 1: Dose 180μg/kg | Part 1: Dose 210μg/kg | Part 1: Dose 240μg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Clinically Significant Physical Examination Results
Description: Clinical significance was determined by the investigator.
Time Frame: Day 1 to end of trial, a maximum of 168 days (+ 30 days)
Population: This analysis was planned but data was not collected as the study was terminated due to safety reasons.
Arm/Group | Part 1: Dose 30μg/kg | Part 1: Dose 60μg/kg | Part 1: Dose 120μg/kg | Part 1: Dose 150μg/kg | Part 1: Dose 180μg/kg | Part 1: Dose 210μg/kg | Part 1: Dose 240μg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants Who Experience a Clinically Significant Change in Eastern Cooperative Oncology Group (ECOG) Performance Status
Description: Performance status was assessed using the ECOG performance status grades. These range between Grade 0 (fully active) and Grade 5 (dead). Clinical significance was determined by the investigator.
Time Frame: Day 1 to end of trial, a maximum of 168 days (+ 30 days)
Population: This analysis was planned but data was not collected as the study was terminated due to safety reasons.
Arm/Group | Part 1: Dose 30μg/kg | Part 1: Dose 60μg/kg | Part 1: Dose 120μg/kg | Part 1: Dose 150μg/kg | Part 1: Dose 180μg/kg | Part 1: Dose 210μg/kg | Part 1: Dose 240μg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Participants With Clinically Significant Vital Signs
Description: Vital sign measurements include arterial blood pressure, heart rate, respiratory rate, and body temperature. Clinical significance was determined by the investigator.
Time Frame: Day 1 to end of trial, a maximum of 168 days (+ 30 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Dose 30μg/kg | Part 1: Dose 60μg/kg | Part 1: Dose 120μg/kg | Part 1: Dose 150μg/kg | Part 1: Dose 180μg/kg | Part 1: Dose 210μg/kg | Part 1: Dose 240μg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 5 | 4 | 3 | 3
Participants | 0 | 0 | 1 | 1 | 0 | 2 | 0

9. Primary Outcome: Number of Participants Who Experience Clinically Significant Electrocardiogram (ECG) Results
Description: Standard 12-lead ECG's will be used. Clinical significance was determined by the investigator.
Time Frame: Day 1 to end of trial, a maximum of 168 days (+ 30 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Dose 30μg/kg | Part 1: Dose 60μg/kg | Part 1: Dose 120μg/kg | Part 1: Dose 150μg/kg | Part 1: Dose 180μg/kg | Part 1: Dose 210μg/kg | Part 1: Dose 240μg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 5 | 4 | 3 | 3
Participants | 0 | 0 | 1 | 0 | 1 | 0 | 0

10. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR was defined as the number of participants with a best overall response of Complete Response (CR) or Partial Response (PR) at the time each participant discontinues ADCT-502. Analysis will be determined by the investigator per Response Evaluation In Solid Criteria (RECIST) version 1.1 criteria: partial response is when there is a decrease in sum of target disease ≥ 30%, and complete response is when all lesions have disappeared or all lesions have disappeared and all nodal disease is < 10 mm each.
Time Frame: Screening, day 1 of cycle 3 and cycle 5, then every 4 cycles, approximately every 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Dose 30μg/kg | Part 1: Dose 60μg/kg | Part 1: Dose 120μg/kg | Part 1: Dose 150μg/kg | Part 1: Dose 180μg/kg | Part 1: Dose 210μg/kg | Part 1: Dose 240μg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 5 | 4 | 3 | 3
Participants
  Complete Response | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 0 | 1 | 0 | 0 | 0

11. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the number of participants with a best overall response of Complete Response (CR) or Partial Response (PR), or Stable Disease (SD). Analysis will be determined by the investigator per Response Evaluation In Solid Criteria (RECIST) version 1.1 criteria: stable disease is when the change is > -30% and ≤ 20%, partial response is when there is a decrease in sum of target disease ≥ 30%, and complete response is when all lesions have disappeared or all lesions have disappeared and all nodal disease is < 10 mm each.
Time Frame: Screening, day 1 of cycle 3 and cycle 5, then every 4 cycles, approximately every 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Dose 30μg/kg | Part 1: Dose 60μg/kg | Part 1: Dose 120μg/kg | Part 1: Dose 150μg/kg | Part 1: Dose 180μg/kg | Part 1: Dose 210μg/kg | Part 1: Dose 240μg/kg
Number analyzed (Participants) | 2 | 2 | 2 | 5 | 4 | 3 | 3
Participants
  Complete Response | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Partial Response | 0 | 0 | 0 | 1 | 0 | 0 | 0
  Stable Disease | 2 | 1 | 0 | 4 | 2 | 2 | 0

12. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined among responders (CR or PR) as the time from the earliest date of first response until the first date of either disease progression or death due to any cause.
Time Frame: Screening, day 1 of cycle 3 and cycle 5, then every 4 cycles, approximately every 12 weeks
Population: This analysis was planned but data was not collected as the study was terminated due to safety reasons.
Groups:
- Part 1: Dose 210μg/kg: Dose-escalation part of the study. Participants received ADCT-502 as a 210μg/kg dose.
Arm/Group | Part 1: Dose 30μg/kg | Part 1: Dose 60μg/kg | Part 1: Dose 120μg/kg | Part 1: Dose 150μg/kg | Part 1: Dose 180μg/kg | Part 1: Dose 210μg/kg | Part 1: Dose 240μg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was defined among the efficacy population as the time from first dose of study drug until the first date of either disease progression or death due to any cause.
Time Frame: Screening, day 1 of cycle 3 and cycle 5, then every 4 cycles, approximately every 12 weeks
Population: This analysis was planned but data was not collected as the study was terminated due to safety reasons.
Groups:
- Part 1: Dose 150μg/kg: Dose-escalation part of the study. Participants received ADCT-502 as a 150μg/kg dose.
- Part 1: Dose 180μg/kg: Dose-escalation part of the study. Participants received ADCT-502 as a 180μg/kg dose.
Arm/Group | Part 1: Dose 30μg/kg | Part 1: Dose 60μg/kg | Part 1: Dose 120μg/kg | Part 1: Dose 150μg/kg | Part 1: Dose 180μg/kg | Part 1: Dose 210μg/kg | Part 1: Dose 240μg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Overall Survival (OS)
Description: Median OS was defined as the time from the beginning of study drug treatment until death due to any cause.
Time Frame: Screening, day 1 of cycle 3 and cycle 5, then every 4 cycles, approximately every 12 weeks
Population: This analysis was planned but data was not collected as the study was terminated due to safety reasons.
Arm/Group | Part 1: Dose 30μg/kg | Part 1: Dose 60μg/kg | Part 1: Dose 120μg/kg | Part 1: Dose 150μg/kg | Part 1: Dose 180μg/kg | Part 1: Dose 210μg/kg | Part 1: Dose 240μg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) of ADCT-502 (Total Antibody)
Time Frame: Before infusion, End of Infusion, and 1, 3, 6, 24, 48, 96, 168 and 336 hours post infusion for Cycle 1 & 2. Before infusion and end of infusion of Cycle 3 to disease progression, and 30 days and 12 weeks after last dose
Population: This analysis was planned but data was not collected as the study was terminated due to safety reasons.
Arm/Group | Part 1: Dose 30μg/kg | Part 1: Dose 60μg/kg | Part 1: Dose 120μg/kg | Part 1: Dose 150μg/kg | Part 1: Dose 180μg/kg | Part 1: Dose 210μg/kg | Part 1: Dose 240μg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Area Under the Plasma Concentration Time Curve (AUC) of Drug To-antibody Ratio [DAR] ≥0
Time Frame: as for outcome 15
Population: This analysis was planned but data was not collected as the study was terminated due to safety reasons.
Arm/Group | Part 1: Dose 30μg/kg | Part 1: Dose 60μg/kg | Part 1: Dose 120μg/kg | Part 1: Dose 150μg/kg | Part 1: Dose 180μg/kg | Part 1: Dose 210μg/kg | Part 1: Dose 240μg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) of PBD-conjugated Antibody (DAR ≥1)
Time Frame: as for outcome 15
Population: This analysis was planned but data was not collected as the study was terminated due to safety reasons.
Arm/Group | Part 1: Dose 30μg/kg | Part 1: Dose 60μg/kg | Part 1: Dose 120μg/kg | Part 1: Dose 150μg/kg | Part 1: Dose 180μg/kg | Part 1: Dose 210μg/kg | Part 1: Dose 240μg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

18. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve (AUC) of Free Warhead SG3199
Time Frame: as for outcome 15
Population: This analysis was planned but data was not collected as the study was terminated due to safety reasons.
Arm/Group | Part 1: Dose 30μg/kg | Part 1: Dose 60μg/kg | Part 1: Dose 120μg/kg | Part 1: Dose 150μg/kg | Part 1: Dose 180μg/kg | Part 1: Dose 210μg/kg | Part 1: Dose 240μg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for ADCT-502 (Total Antibody)
Time Frame: as for outcome 15
Population: This analysis was planned but data was not collected as the study was terminated due to safety reasons.
Arm/Group | Part 1: Dose 30μg/kg | Part 1: Dose 60μg/kg | Part 1: Dose 120μg/kg | Part 1: Dose 150μg/kg | Part 1: Dose 180μg/kg | Part 1: Dose 210μg/kg | Part 1: Dose 240μg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

20. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for Drug To-antibody Ratio [DAR] ≥0
Time Frame: as for outcome 15
Population: This analysis was planned but data was not collected as the study was terminated due to safety reasons.
Arm/Group | Part 1: Dose 30μg/kg | Part 1: Dose 60μg/kg | Part 1: Dose 120μg/kg | Part 1: Dose 150μg/kg | Part 1: Dose 180μg/kg | Part 1: Dose 210μg/kg | Part 1: Dose 240μg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

21. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for PBD-conjugated Antibody (DAR ≥1)
Time Frame: as for outcome 15
Population: This analysis was planned but data was not collected as the study was terminated due to safety reasons.
Arm/Group | Part 1: Dose 30μg/kg | Part 1: Dose 60μg/kg | Part 1: Dose 120μg/kg | Part 1: Dose 150μg/kg | Part 1: Dose 180μg/kg | Part 1: Dose 210μg/kg | Part 1: Dose 240μg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) for Free Warhead SG3199
Time Frame: as for outcome 15
Population: This analysis was planned but data was not collected as the study was terminated due to safety reasons.
Arm/Group | Part 1: Dose 30μg/kg | Part 1: Dose 60μg/kg | Part 1: Dose 120μg/kg | Part 1: Dose 150μg/kg | Part 1: Dose 180μg/kg | Part 1: Dose 210μg/kg | Part 1: Dose 240μg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

23. Secondary Outcome: Time to Reach the Maximum Plasma Concentration (Tmax) for ADCT-502 (Total Antibody)
Time Frame: as for outcome 15
Population: This analysis was planned but data was not collected as the study was terminated due to safety reasons.
Arm/Group | Part 1: Dose 30μg/kg | Part 1: Dose 60μg/kg | Part 1: Dose 120μg/kg | Part 1: Dose 150μg/kg | Part 1: Dose 180μg/kg | Part 1: Dose 210μg/kg | Part 1: Dose 240μg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

24. Secondary Outcome: Time to Reach the Maximum Plasma Concentration (Tmax) for Drug To-antibody Ratio [DAR] ≥0)
Time Frame: as for outcome 15
Population: This analysis was planned but data was not collected as the study was terminated due to safety reasons.
Arm/Group | Part 1: Dose 30μg/kg | Part 1: Dose 60μg/kg | Part 1: Dose 120μg/kg | Part 1: Dose 150μg/kg | Part 1: Dose 180μg/kg | Part 1: Dose 210μg/kg | Part 1: Dose 240μg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

25. Secondary Outcome: Time to Reach the Maximum Plasma Concentration (Tmax) for PBD-conjugated Antibody (DAR ≥1)
Time Frame: as for outcome 15
Population: This analysis was planned but data was not collected as the study was terminated due to safety reasons.
Arm/Group | Part 1: Dose 30μg/kg | Part 1: Dose 60μg/kg | Part 1: Dose 120μg/kg | Part 1: Dose 150μg/kg | Part 1: Dose 180μg/kg | Part 1: Dose 210μg/kg | Part 1: Dose 240μg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

26. Secondary Outcome: Time to Reach the Maximum Plasma Concentration (Tmax) for Free Warhead SG3199
Time Frame: as for outcome 15
Population: This analysis was planned but data was not collected as the study was terminated due to safety reasons.
Arm/Group | Part 1: Dose 30μg/kg | Part 1: Dose 60μg/kg | Part 1: Dose 120μg/kg | Part 1: Dose 150μg/kg | Part 1: Dose 180μg/kg | Part 1: Dose 210μg/kg | Part 1: Dose 240μg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

27. Secondary Outcome: Anti-drug Antibody (ADA) Titers to ADCT-502
Time Frame: Blood sample collection before start of infusion in Cycles 1 and 2, and on Day 1 starting with Cycle 3 until disease progression, 30 days and 12 weeks after last dose
Population: This analysis was planned but data was not collected as the study was terminated due to safety reasons.
Arm/Group | Part 1: Dose 30μg/kg | Part 1: Dose 60μg/kg | Part 1: Dose 120μg/kg | Part 1: Dose 150μg/kg | Part 1: Dose 180μg/kg | Part 1: Dose 210μg/kg | Part 1: Dose 240μg/kg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to end of trial, a maximum of 168 days (+ 30 days)
Arm/Group | Part 1: Dose 30μg/kg | Part 1: Dose 60μg/kg | Part 1: Dose 120μg/kg | Part 1: Dose 150μg/kg | Part 1: Dose 180μg/kg | Part 1: Dose 210μg/kg | Part 1: Dose 240μg/kg
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/5 | 0/4 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 1/2 | 0/2 | 2/5 | 1/4 | 2/3 | 1/3
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 2/2 | 5/5 | 4/4 | 3/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Dose 30μg/kg (N=2) | Part 1: Dose 60μg/kg (N=2) | Part 1: Dose 120μg/kg (N=2) | Part 1: Dose 150μg/kg (N=5) | Part 1: Dose 180μg/kg (N=4) | Part 1: Dose 210μg/kg (N=3) | Part 1: Dose 240μg/kg (N=3)
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Klebsiella infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Dose 30μg/kg (N=2) | Part 1: Dose 60μg/kg (N=2) | Part 1: Dose 120μg/kg (N=2) | Part 1: Dose 150μg/kg (N=5) | Part 1: Dose 180μg/kg (N=4) | Part 1: Dose 210μg/kg (N=3) | Part 1: Dose 240μg/kg (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Photophobia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 2 | 2 | 0 | 2 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lip ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 1 | 5 | 2 | 2 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 3 | 1 | 1 | 2
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 3 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Body tinea (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Candida infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hordeolum (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Klebsiella infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Weight increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 3 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Bone disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 3 | 1 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 2 | 1 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 3 | 0 | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 2 | 1 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI can publish after first multi-site publication, or if no multi-site publication is made within 18 months of study completion/termination. The only disclosure restriction on the PI is the sponsor can review results comms. prior to public release and can embargo comms. regarding trial results for a period that is more than 60 but less than or equal to 180 days from the time submitted to sponsor for review. The sponsor can't require changes to the communication and can't extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2017-08-17): https://cdn.clinicaltrials.gov/large-docs/00/NCT03125200/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-05): https://cdn.clinicaltrials.gov/large-docs/00/NCT03125200/SAP_001.pdf